CLINICAL TRIAL: NCT04757207
Title: The Effect of Pandemia on Making Exercise In University Students of Turkey
Brief Title: Pandemia And Exercise in Turkey in University Students of Turkey
Status: Completed | Type: Observational
Sponsor: GULIN FINDIKOGLU (Other)
Responsible Party: Sponsor-Investigator, GULIN FINDIKOGLU, Assoc Proffessor, MD, PhD, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: 60116787-020/76132
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Sedentary Behavior; Covid19
MeSH Terms: conditions — Sedentary Behavior; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — International Physical Activity Questionnaire (short form)

SUMMARY:
The aim of this study is to determine to what extent university students' physical activities are affected by staying at home during the pandemia.

DETAILED DESCRIPTION:
The aim of our study is to determine to what extent university students' physical activities are affected by staying at home during the pandemia considering that they spend hours working by a computer. The state of physical inactivities will be questioned by an online survey for Inernational Physical Activity Questionnaire (short form). Then average energy expenditure following stepping and/or exercise will be asked from health application of mobile phones.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student
* Having sufficient device infrastructure (cell phone or computer) to access the electronic survey

Exclusion Criteria:

* Entering incorrect numbers for answers
* Those who have a disease / disability that prevents them from walking and exercising

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Being a university student
  * Having sufficient devices (cell phone or computer) to access the electronic survey
Sampling Method: Non-Probability Sample
Enrollment: 5474 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Score (short form) MEt-min/week | an average of 2 months, through study completion.
  International Physical Activity Score (short form) during pandemia. Higher scores indicate better physical activity status. There is no strict range.

SECONDARY OUTCOMES:
Energy expenditure while stepping | an average of 2 months, through study completion.
  Energy expenditure while stepping during pandemia and before pandemia (Kcal)
Energy expenditure while exercising | an average of 2 months, through study completion.
  Energy expenditure while exercising during pandemia and before pandemia (Kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No